CLINICAL TRIAL: NCT01176253
Title: Detection of Human Beta Cell Death in T1DM by Methylation Specific PCR
Brief Title: Detection of Human Beta Cell Death in Type 1 Diabetes Mellitus (T1DM) by Methylation Specific Polymerase Chain Reaction (PCR)
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08078
Record Dates: First submitted 2010-08-04; First posted 2010-08-05 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type I DM
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 25 newly diagnosed Type 1 diabetics: 25 newly diagnosed Type 1 diabetics within onset of symptoms
  Interventions: Procedure: Blood draw
- 25 healthy volunteers: 25 healthy volunteers (age & sex matched)
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — Blood draw for Type I DM patients will be taken every 4 weeks for 1 year post diagnosis/healthy volunteers will have 1 blood draw

SUMMARY:
To investigate the use of methylation-specific PCR (MSP) assays to detect human beta cell-specific gene methylation patterns in serial blood samples drawn from newly diagnosed Type 1 diabetics.

DETAILED DESCRIPTION:
The study will follow 25 newly diagnosed type 1 diabetic patients from the onset of symptoms to one year post-diagnosis. A total of 11 fasting blood draws will be taken, the first near the time of diabetes diagnosis, then 2 weeks later, monthly for the next 6 months, and every other month until 12 months. Each blood sample will be evaluated by the MSP assay, as well as for measurement of fasting plasma glucose, HbA1c, c-peptide, and autoantibodies. The study will also need 25 healthy volunteers to help us match some DNA markers needed for this data. Healthy volunteers will be se=matched healthy individuals who have one blood sample drawn.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Age > 18 years of age,
* Otherwise healthy individuals with no cancer and not pregnant.

Type 1DM:

* Newly diagnosed type I diabetes,
* Age > 18 years of age,
* Otherwise healthy individuals with no severe complications, no cancer, not pregnant,
* Willing and able to comply with the scheduled visits to the clinic for blood sampling,
* Remain under the continuing care of an Endocrinologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type I Diabetic, newly diagnosed, >18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2009-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Develop sensitive, specific, and quantitative methylation- specific PCR assays for the detection of human beta cell-specific DNA methylation patterns cells and the onset of metabolic dysregulation. | 1 year post diagnosis
Use the assays to detect beta cell destruction throughout the early time-course of type 1 diabetes mellitus | 1 year post diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ferreri, Ph.D., Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope National Medical Center-Department of Diabetes, Endocrinology, & Metabolism, Duarte, California
  - Loma Linda Medical Center, Loma Linda, California

REFERENCES:
- [Background] Lo YM. Circulating nucleic acids in plasma and serum: an overview. Ann N Y Acad Sci. 2001 Sep;945:1-7. doi: 10.1111/j.1749-6632.2001.tb03858.x. PMID 11708462
- [Background] Schutz E, Urnovitz HB, Iakoubov L, Schulz-Schaeffer W, Wemheuer W, Brenig B. Bov-tA short interspersed nucleotide element sequences in circulating nucleic acids from sera of cattle with bovine spongiform encephalopathy (BSE) and sera of cattle exposed to BSE. Clin Diagn Lab Immunol. 2005 Jul;12(7):814-20. doi: 10.1128/CDLI.12.7.814-820.2005. PMID 16002628
- [Background] Tong YK, Lo YM. Diagnostic developments involving cell-free (circulating) nucleic acids. Clin Chim Acta. 2006 Jan;363(1-2):187-96. doi: 10.1016/j.cccn.2005.05.048. Epub 2005 Aug 26. PMID 16126188
- [Background] Galm O, Herman JG. Methylation-specific polymerase chain reaction. Methods Mol Med. 2005;113:279-91. doi: 10.1385/1-59259-916-8:279. PMID 15968111
- [Background] Koike H, Ichikawa D, Ikoma H, Otsuji E, Kitamura K, Yamagishi H. Comparison of methylation-specific polymerase chain reaction (MSP) with reverse transcriptase-polymerase chain reaction (RT-PCR) in peripheral blood of gastric cancer patients. J Surg Oncol. 2004 Sep 15;87(4):182-6. doi: 10.1002/jso.20106. PMID 15334633
- [Background] Liu Q, Sommer SS. Detection of extremely rare alleles by bidirectional pyrophosphorolysis-activated polymerization allele-specific amplification (Bi-PAP-A): measurement of mutation load in mammalian tissues. Biotechniques. 2004 Jan;36(1):156-66. doi: 10.2144/04361DD03. PMID 14740499
- [Background] Gierl MS, Karoulias N, Wende H, Strehle M, Birchmeier C. The zinc-finger factor Insm1 (IA-1) is essential for the development of pancreatic beta cells and intestinal endocrine cells. Genes Dev. 2006 Sep 1;20(17):2465-78. doi: 10.1101/gad.381806. PMID 16951258
- [Background] Wang J, Cortina G, Wu SV, Tran R, Cho JH, Tsai MJ, Bailey TJ, Jamrich M, Ament ME, Treem WR, Hill ID, Vargas JH, Gershman G, Farmer DG, Reyen L, Martin MG. Mutant neurogenin-3 in congenital malabsorptive diarrhea. N Engl J Med. 2006 Jul 20;355(3):270-80. doi: 10.1056/NEJMoa054288. PMID 16855267